CLINICAL TRIAL: NCT03795350
Title: Open Label, Uncontrolled, Non-randomized, Single Dose, Scintigraphic Study to Investigate Lung Deposition of Inhaled 99mTc Radiolabelled TRIMBOW® pMDI in Healthy Volunteers, Asthmatic and COPD Patients
Brief Title: Lung Deposition of TRIMBOW® pMDI in Healthy Volunteers, Asthmatic and COPD Patients
Acronym: STORM
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: In light of the cessation of non-essential clinical activities at CPU due to the COVID-19 pandemic, the sponsor has determined to terminate the study early.
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLI-05993AA1-20; 2017-005030-29 (EudraCT Number)
Record Dates: First submitted 2018-12-18; First posted 2019-01-07 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Chronic Obstructive Pulmonary Disease; Asthma
Keywords: Lung deposition; Gamma scintigraphy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TRIMBOW (Experimental): Experimental: BDP/FF/GB
  4 puffs of 99mTc Radiolabelled Beclometasone dipropionate/Formoterol Fumarate/Glycopyrronium Bromide administered via pMDI
  Interventions: Drug: Beclometasone dipropionate Formoterol Fumarate Glycopyrronium Bromide

INTERVENTIONS:
Drug: Beclometasone dipropionate Formoterol Fumarate Glycopyrronium Bromide — single inhalation of 99mTc radiolabelled TRIMBOW pMDI (4 puffs for a total dose of 400mcg BDP, 24mcg FF, 50 mcg GB)

SUMMARY:
The purpose of this study is to investigate the lung deposition and distribution pattern of TRIMBOW using a Gamma-scintigraphic technique after inhalation of a single dose of 99mTc radiolabelled TRIMBOW administered via pMDI in healthy volunteers, asthmatic and COPD patients

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for all subjects:

1. Subject's written informed consent obtained prior to any study-related procedure;
2. Ability to understand the study procedures, the risks involved and ability to demonstrate correct use of the inhaler using the AIM™ (Aerosol Inhalation Monitor) Vitalograph®
3. Body Mass Index (BMI) between 18 and 32 kg/m2 extremes inclusive;
4. Good physical status, determined on the basis of the medical history and a general clinical examination, at screening;
5. Vital signs within normal limits: Diastolic BP 40-90 mmHg, Systolic BP 90-140 mmHg or 90-160 mmHg if >45 yrs
6. Males fulfilling one of the following criteria:

   1. Males with non-pregnant Women of childbearing potential (WOCBP) partners: they and/or their partner of childbearing potential must be willing to use a highly effective birth control method in addition to the male condom from the signature of the informed consent and until 90 days after the follow-up visit. Subjects must not donate sperm during the study and for 90 days after the follow-up visit or
   2. Males with pregnant WOCBP partner: they must be willing to use male contraception (condom) from the signature of the informed consent and until 90 days after the follow-up visit. Subjects must not donate sperm during the study and for 90 days after the follow-up visit or
   3. Non-fertile male subjects (contraception is not required in this case) or
   4. Males with partner not of childbearing potential (contraception is not required in this case).
7. WOCBP fulfilling one of the following criteria:

   1. WOCBP with fertile male partners: they and/or their partner must be willing to use a highly effective birth control method with low user dependency from the signature of the informed consent and until 30 days after the follow-up visit or
   2. WOCBP with non-fertile male partners (contraception is not required in this case).
8. Females of non-childbearing potential defined as physiologically incapable of becoming pregnant (i.e. post-menopausal or permanently sterile). Tubal ligation or partial surgical interventions are not acceptable. If indicated, as per investigator's request, post-menopausal status may be confirmed by follicle-stimulating hormone levels (according to local laboratory ranges)
9. 12 -lead digitised Electrocardiogram (12-lead ECG) considered as normal at screening and at Day -1

Additional Criteria only for Healthy Volunteers and Asthmatic patients:

1. Male and female subjects aged 28-55 years inclusive;
2. Non- or ex-smokers who smoked < 5 pack years (pack-years = the number of cigarette packs per day times the number of years) and stopped smoking > 6 months prior to screening;

Additional Inclusion Criteria only for Healthy Volunteers:

1. Lung function measurements within normal limits at screening: FEV1 equal to or more than 80% of predicted

Additional Inclusion Criteria only for Asthmatic patients:

1. Diagnosis of asthma: Established diagnosis of permanent asthma for at least 12 months according to GINA guidelines
2. Patients with a pre-bronchodilator 60%≤ FEV1 < 80% of the predicted normal value
3. Patients with a documented reversibility defined as an increase ≥ 12% and 200mL over baseline within 30 min after inhalation of 400µg salbutamol pMDI

Additional Inclusion Criteria only for COPD patients:

1. Male and female patients aged 40-80 years inclusive
2. A smoking history of at least 10 pack-years
3. Current or ex-smokers are eligible.
4. Established diagnosis of COPD
5. A post-bronchodilator FEV1 ≤ 50% of the predicted normal value and a post-bronchodilator FEV1/FVC < 0.7 10-15 minutes after 4 puffs (4x100 µg) of Salbutamol pMDI.

Exclusion Criteria:

Inclusion criteria for all subjects:

1. Pregnant or lactating women;
2. Clinically relevant and uncontrolled respiratory, cardiac, hepatic, gastrointestinal, renal, endocrine, metabolic, neurologic, or psychiatric disorders
3. Clinically relevant abnormal laboratory values at screening suggesting an unknown disease and requiring further clinical investigation
4. Subjects with medical diagnosis of narrow-angle glaucoma, prostatic hypertrophy or bladder neck obstruction
5. Positive HIV1 or HIV2 serology at screening
6. Blood donation or blood loss less than 2 months prior screening
7. Participation to another clinical trial where investigational drug was received and last investigations were performed less than 90 days prior to screening;
8. Documented history of alcohol abuse within 12 months prior to screening or a positive alcohol breath test
9. Documented history of drug abuse within 12 months prior to screening
10. Positive results from the Hepatitis serology which indicates acute or chronic Hepatitis B or Hepatitis C at screening
11. Subjects who have cardiovascular condition such as, but not limited to unstable ischemic heart disease, NYHA Class III/IV left ventricular failure, acute ischemic heart disease in the last year prior to study screening, which may impact the safety of the subject or the evaluation of the result of the study according to the Investigator's judgment
12. Unsuitable veins for repeated venepuncture/cannulation
13. Intake of non-permitted concomitant medications in the predefined period prior to screening
14. Radiation exposure, including that from the present study, in the last 12 months
15. Known intolerance/hypersensitivity or contra-indication to treatment

Additional exclusion Criteria only for Healthy volunteers and Asthmatic patients:

1. Positive urine test for cotinine at screening or prior Day 1
2. Current use of any nicotine or nicotine replacement product

Additional exclusion criteria only for Asthmatic and COPD patients:

1. Use of systemic corticosteroids medication within 4 weeks prior to the screening or slow release corticosteroids within 12 weeks before the screening or prior Day 1
2. A diagnosis of lung cancer or a history of lung cancer
3. A history of lung volume reduction surgery
4. Lower respiratory tract infection that requires use of antibiotics

Additional exclusion Criteria only for Healthy volunteers:

1. Subjects with history of breathing problems

Additional exclusion Criteria only for Asthmatic patients:

1. History of near fatal asthma, hospitalization for asthma in intensive care unit
2. Any change in dose, schedule or formulation in the treatment of asthma in the 4 weeks prior to the screening visit or prior Day 1
3. Non-persistent asthma:
4. Treatment with chronic systemic corticosteroids or anti IgE or other monoclonal antibodies
5. Known respiratory disorders other than asthma

Additional exclusion Criteria only for COPD patients:

1. Any change in dose, schedule or formulation in the treatment for COPD in the 4 weeks prior to the screening
2. A concurrent diagnosis of asthma, in the opinion of the investigator
3. Known respiratory disorder other than COPD that in the Investigator's opinion would affect efficacy and safety evaluation or place the patient at risk.
4. Oxygen therapy: patients requiring long term (at least 12 hours daily) oxygen therapy for chronic hypoxemia.
5. Change in dose or type of any medications for COPD within 4 weeks prior to the screening visit.

Ages: 28 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2020-04-03 (Actual); Study Completion 2020-04-03 (Actual)

PRIMARY OUTCOMES:
intrapulmonary lung deposition | immediately after dosing
  calculated using individual Gamma camera images

SECONDARY OUTCOMES:
Intrapulmonary lung distribution of deposition: C/P ratio | immediately after dosing
extrathoracic deposition | immediately after dosing
amount of exhaled drug | immediately after dosing
TRIMBOW pharmacokinetics - (AUC0-t) | up to 24 hours post dose
  Area Under plasma Concentration from 0 to last quantifiable concentration (AUC0-t) for BDP, B17MP, FF and GB
lung function assessment - FEV1, FVC, FEV1/FVC, FEF25%, FEF50%, FEF75% | up to 24 hours post dose
  FEV1, FVC, FEV1/FVC, FEF25%, FEF50%, FEF75%
TRIMBOW pharmacokinetics - (AUC0-30) | up to 24 hours post dose
  area under plasma concentration from 0 to 30 min (AUC0-30) for B17MP, FF and GB
TRIMBOW pharmacokinetics - (Cmax) | up to 24 hours post dose
  Maximum plasma concentration (Cmax) for BDP, B17MP, FF and GB
TRIMBOW - (tmax) | up to 24 hours post dose
  time of the maximum plasma concentration (tmax) for BDP, B17MP, FF and GB
TRIMBOW pharmacokinetics - (AUC0-∞) | up to 24 hours post dose
  area under curve extrapolated to infinity (AUC0-∞) for B17MP, FF and GB
TRIMBOW pharmacokinetics - (t1/2) | up to 24 hours post dose
  terminal half-life (t1/2) for B17MP, FF and GB

CONTACTS AND LOCATIONS:
Locations (1):
- Simbec Research Ltd, Merthyr Tydfil, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Usmani OS, Baldi S, Warren S, Panni I, Girardello L, Rony F, Taylor G, DeBacker W, Georges G. Lung Deposition of Inhaled Extrafine Beclomethasone Dipropionate/Formoterol Fumarate/Glycopyrronium Bromide in Healthy Volunteers and Asthma: The STORM Study. J Aerosol Med Pulm Drug Deliv. 2022 Aug;35(4):179-185. doi: 10.1089/jamp.2021.0046. Epub 2022 Feb 4. PMID 35128939